CLINICAL TRIAL: NCT06289842
Title: Efficacy of Accelerated Theta Burst Stimulation for Treatment of Suicidality in Patients With Unipolar and Bipolar Depression
Brief Title: Accelerated Theta Burst Stimulation for Treatment of Suicidality in Depressed Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Medhat Bassiony, Professor of Psychiatry, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZU-IRB #9697
Record Dates: First submitted 2024-02-24; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Suicide and Depression
MeSH Terms: conditions — Suicide; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unipolar depressed patients with suicidality (Active Comparator): The participants will receive iTBS (intermittent theta burst stimulation) to the left dorsolateral prefrontal cortex (LDLPFC) determined using Beam method for 1800 pulses with an intertreatment interval of fifty minutes. Stimulation was at 120% of resting motor threshold. Patients received ten sessions every day for five consecutive days for a total of fifty sessions (90,000 pulses).
  Interventions: Device: Transcranial Magnetic Stimulation MagPro R30 with the MCF-B70 figure-of-eight coil (MagVenture, Denmark)
- Bipolar depressed patients with suicidality (Active Comparator): The participants will receive iTBS (intermittent theta burst stimulation) to the left dorsolateral prefrontal cortex (LDLPFC) determined using Beam method for 1800 pulses with an intertreatment interval of fifty minutes. Stimulation was at 120% of resting motor threshold. Patients received ten sessions every day for five consecutive days for a total of fifty sessions (90,000 pulses).
  Interventions: Device: Transcranial Magnetic Stimulation MagPro R30 with the MCF-B70 figure-of-eight coil (MagVenture, Denmark)

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation MagPro R30 with the MCF-B70 figure-of-eight coil (MagVenture, Denmark) — TMS Therapy System with Theta Burst Stimulation

SUMMARY:
The objective of this study is to investigate efficacy of accelerated theta burst stimulation (TBS) in suicidal reduction in patients with unipolar and bipolar depression

DETAILED DESCRIPTION:
Introduction:

Depression is the leading cause of disability worldwide and is associated with increased suicide risk, morbidity and mortality.(Sousa et al .,2022).

In severe cases, depression can result in suicide and approximately 800,000 suicides occur each year (Lepine et al.,2011). Rates of completed suicide are also high, varying from 10 to 19% (Goodwin et al., 1990). Lifetime rates of attempted suicide in bipolar depression range (26-29%) and (14-16%) in unipolar depression disorder (Chen et al., 1996).

The general recommendation to reduce suicide risk is the effective treatment of the underlying depressive disorder, with medications and psychosocial interventions (Jacobs et al., 2010). However, there exist several difficulties. Neither antidepressants nor psychotherapy work fast enough for reduction of suicidal ideation.

Beside pharmacotherapy and psychotherapy brain stimulation methods have gained increasing relevance in the treatment of depression during the last decades (Baeken et al.,2019).

Repetitive transcranial magnetic stimulation (rTMS) therapy is a noninvasive neurostimulation treatment that has been adopted as a first-line treatment for pharmacotherapy-resistant major depressive disorder (MDD) (Milev et al., 2016).

Despite this growing evidence base supporting (iTBS) in the treatment of MDD, evidence for its efficacy in the treatment of suicidality as a primary outcome in both unipolar and bipolar depressive patients is still lacking.

Hypothesis We assume that accelerated TBS is effective in treatment of suicidality as well as depressive symptoms in both unipolar and bipolar patients.

Aim This study aims to reduce morbidity and mortality of unipolar and bipolar depressive patients and to improve overall functioning.

Objectives

1. To investigate efficacy of accelerated TBS in suicidal reduction as primary outcome in patients with unipolar and bipolar depression.
2. To compare efficacy of accelerated TBS in reduction of severity of depressive symptoms in unipolar and bipolar disorder as well as response and remission rates.
3. To investigate association between the reduction of suicidality and the reduction of depressive symptoms

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major depressive episode as a part of MDD or bipolar (I or II) disorder and confirmed by Structured Clinical Interview for DSM-IV-TR Axis I Disorders (SCID-I). (First & Gibbon.,2004 ).
* Meeting the severe depression cutoff for MADRS (>/=35) at baseline visit.
* Meeting the severe depression cutoff for BDI-II (>/=30) at baseline visit.
* Presence of suicidal ideation and/or behavior (confirmed with Columbia Scale for the Rating of Suicide Severity (C-SSRS)
* Adults (Age 19 years or older )
* Right handedness
* Both genders
* Able to provide informed consent to participate in the study
* Participants were required to have been taking a stable pharmacological regimen for 2 weeks before screening.
* Pass the TMS adult safety screening (TASS) questionnaire

Exclusion Criteria

* Current substance use disorder during the past 3 months
* Current psychotic disorder or symptoms
* Presence of dementia
* Presence of major medical illness, for example metastatic cancer, end stage renal disease
* Inability to verify contact information.
* Presence of any clinically significant neurological disorder, including organic brain disease, epilepsy, stroke, brain lesions, previous neurosurgery, or personal history of head trauma that resulted in loss of consciousness for > 5 minutes and retrograde amnesia for > 30 minutes
* Conductive, ferromagnetic or other magnetic sensitive metals that are implanted or are non-removable within 30 cm treatment coil (around the head)
* Presence of hypomanic symptoms (score on Young Mania Rating Scale (YMRS) greater than 12)
* Current severe insomnia (must sleep a minimum of 5 hours the night before stimulation)
* Using lorazepam greater than 2 mg daily (or equivalent) due to the potential to limit rTMS efficacy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in suicidal ideation and behaviors as measured by Columbia Suicide Severity Rating Scale (C-SSRS) | Assessed at baseline (day 0) , post-inpatient treatment completion (day 5) , 1 month ,3 month , 6 month, 9 month and 12 month
  The SI severity scale is composed of five yes=no questions of increasingly severe suicidal thoughts: a wish to be dead (1), non-specific suicidal thoughts (2), suicidal thoughts with a method (3), suicidal intent without specific plan (4), and suicidal intent with specific plan (5).
  This scale was scored from 0 to 5 according to the most severe suicidal ideation endorsed. Higher scores mean worse outcome.
  Suicidal behaviors were assessed dichotomously (yes=no) and include actual suicide attempts, interrupted suicide attempts, aborted suicide attempts, other preparatory acts (e.g., collecting pills, writing suicide note), and non-suicidal self-injury (NSSI).

SECONDARY OUTCOMES:
Change from baseline Montgomery-Åsberg Depression Rating Scale (MADRS) Score | Assessed at baseline (day 0) , post-inpatient treatment completion (day 5) , 1 month ,3 month , 6 month ,9 months and 12 month
  The Montgomery-Åsberg Depression Rating Scale (MADRS), is a ten item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60.

CONTACTS AND LOCATIONS:
Overall Officials: Medhat M Bassiony, Professor, Principal Investigator — Zagazig University
Locations (1):
- Zagazig University, Zagazig, Egypt